CLINICAL TRIAL: NCT05599243
Title: Exploratory Clinical Trial of Safety and Efficacy of Daily Application of Topical Dutasteride in Men With Androgenic Alopecia.
Brief Title: Clinical Trial of Safety and Efficacy of Daily Application of Topical Dutasteride in Men With Androgenic Alopecia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALOSTOP
Record Dates: First submitted 2022-10-03; First posted 2022-10-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Male Androgenetic Alopecia
MeSH Terms: interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental drug (Experimental): 0.15% w/w dutasteride topical O/W emulsion.
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator): vehicle (excipients)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dutasteride — The application will be made locally (spray for topical application on the scalp) Application: 1 mL (6 sprays) once a day. Each 1mL of formulation has approximately 1.5mg of Dutasteride (more precisely it would be 1.4835mg when considering density).
  Arms: experimental drug
Other: Placebo — Vehicle excipient
  Arms: Placebo

SUMMARY:
Alopecia is a disorder that involves the loss of hair from the body. The causes of hair loss can be multiple, but in all cases this loss causes a lot of discomfort to patients for aesthetic and psychological reasons, especially in the female population.This study is going to focus on the topical use of dutasteride in the treatment of men with androgenic alopecia using a new formulation, as an emulsion, capable of transporting this drug to the different structures of the pilosebaceous unit.

DETAILED DESCRIPTION:
Alopecia is a disorder that involves the loss of hair from the body. The causes of hair loss can be multiple, but in all cases this loss causes a lot of discomfort to patients for aesthetic and psychological reasons, especially in the female population. This disorder, although more visible in men, is suffered by both men and women. Recent studies show that the stress experienced by patients with alopecia can be similar or greater than that suffered by a more serious or chronic disease. For all these reasons, alopecia can prefer a social problem without a definitive therapeutic solution.This study is going to focus on the topical use of dutasteride in the treatment of men with androgenic alopecia using a new formulation, as an emulsion, capable of transporting this drug to the different structures of the pilosebaceous unit. The lipid nature of the formulation and the droplet size of between 150-300 nm means that the emulsion drops easily penetrate the hair follicle and accumulate in the sebaceous glands of said follicles.

ELIGIBILITY:
Inclusion Criteria:

* • - Males over 18 years of age, diagnosed with Sinclair grades I-IV androgenic alopecia, who are not currently undergoing any hair treatment and have not undergone any in the last 3 months.

  * - Understand the purpose of the study and be available for frequent visits to the hospital. Sign the informed consent form.
  * - Males with a partner of childbearing age must agree to use a contraceptive method with the partner for the duration of the study.

Exclusion Criteria:

* • - Patients with a history of hypersensitivity to the active ingredient, to other 5-alpha reductase inhibitors.

  * - Patients with severe hepatic insufficiency.
  * - Patients who are currently undergoing capillary treatment or have undergone capillary treatment in the last 3 months.
  * - Patients unable to understand the objective of the study or to give informed consent.
  * - Patients who, in the opinion of the investigator, present any difficulty or situation that would hinder or contraindicate their participation in this study.
  * - Patients with a history of drug addiction and drug addictions.
  * - Patients who are participating in another clinical trial.
  * - Patients whose partner is pregnant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 45 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 7 months
  Local adverse events (AEs) and systemic adverse reactions
  - Hair microbiome analysis

SECONDARY OUTCOMES:
Efficacy in hair loss reduction | 7 months
  Clinical improvement. Standardized photographs will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Muñoz, MD, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No